CLINICAL TRIAL: NCT04879251
Title: The Impact of the COVID-19 Pandemic on Cardiovascular Risk Factors in Patients With Diabetes.
Acronym: ICOVdia
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: 3/IK-FNO/2021
Record Dates: First submitted 2021-05-06; First posted 2021-05-10 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Diabetes Mellitus; Covid19
Keywords: Diabetes Mellitus; COVID 19; LDL hyperlipoproteinemia
MeSH Terms: conditions — Diabetes Mellitus; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The objective of this study is to compare cardiovascular risk factors in patients with diabetes before the start of the pandemic of the COVID 19 (time 1 - T1), after 1 year (time 2 - T2) and 2 years (time 3 - T3) duration. In patients with all types of diabetes, the investigators will compare the value of blood pressure, LDL cholesterol, BMI (body mass index) and glycated haemoglobin in T1, T2 and T3 during outpatient control.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is one of the major risk factors of cardiovascular diseases (CVDs), which are the leading cause of death globally. To reduce overall cardiovascular risk in patients with diabetes, it is necessary, in addition to compensation of diabetes, to reduce other risk factors of cardiovascular diseases. The COVIDs 19 (coronavirus disease of 2019) pandemic has in addition to direct influence (fever, pneumonia, olfactory loss, etc.)1,2 also, a lot of indirect effects. These include psychological effects (long term stress, worries, sadness)3,4,5, increased alcohol consumption, changes in eating habits or decreased physical activity due to restrictions to reduce the spread of the virus in population by government.

The Czech Republic (Central Europe region) is one of the most affected countries in the World by COVID 19 pandemic. By 1st of March 2021, the SARS-COV2 virus infection was proven in the Czech Republic in 1 247 051 thousand people, which is 11.7% of the population (11 627 per 100 000, in the USA 8743/100 000, in the UK 6300/100 000, in the Germany 2879/100 000, France 5379/100 000)6 Due to a long-lasting serious situation, we expect an adverse effect on number of risk factors for CVDs.

The objective of this study is to compare cardiovascular risk factors in patients with diabetes before the start of the pandemic of the COVID 19 (time 1 - T1), after 1 year (time 2 - T2) and 2 years (time 3 - T3) duration. In patients with all types of diabetes, the investigators will compare the value of blood pressure, LDL cholesterol, BMI (body mass index) and glycated haemoglobin in T1, T2 and T3 during outpatient control.

The secondary objective is to evaluate behaviour of patients during COVID 19 pandemic. The investigators will use a questionnaire. It will be anonymous for a more accurate assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Diabetes mellitus of any type
* Planned visit to the outpatient diabetic clinic between 1.4. and 31.7.2021 - T2 (creation of the study group) - University hospital Ostrava, Czech Republic
* Known values of blood pressure, glycated haemoglobin, LDL cholesterol and BMI before the start of the pandemic (1.3.2020), not older than 6 months and no later than 31.3.2020.
* Signed consent to the use of anonymous data for scientific purposes and publications.

Exclusion Criteria:

* failure to meet the criteria for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetes mellitus of any type
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with diabetes who have a worse glycated hemoglobin value (Change from baseline after 1 and 2 year of COVID 19 pandemic) | Baseline values - before the start of COVID 19 pandemic (1.9.2019 - 1.3.2020)- change from baseline after 1 year 1.4. - 31.7. 2020 and after 2 years (1.4.2021-31.7.2022)
  The investigators compare the value of glycated hemoglobin before the start of the COVID 19 pandemic and change from baseline after one year of the pandemic in each participant with diabetes.
Number of patients with diabetes who have a worse LDL cholesterol value (Change from baseline after 1 and 2 year of COVID 19 pandemic) | Baseline values - before the start of COVID 19 pandemic (1.9.2019 - 1.3.2020)- change from baseline after 1 year 1.4. - 31.7. 2020 and after 2 years (1.4.2021-31.7.2022)
  The investigators compare the value of LDL cholesterol before the start of the COVID 19 pandemic and change from baseline after one year of the pandemic in each participant with diabetes.
Number of patients with diabetes who have a higher BMI value (Change from baseline after 1 and 2 year of COVID 19 pandemic) | Baseline values - before the start of COVID 19 pandemic (1.9.2019 - 1.3.2020)- change from baseline after 1 year 1.4. - 31.7. 2020 and after 2 years (1.4.2021-31.7.2022)
  The investigators compare the value of BMI before the start of the COVID 19 pandemic and change from baseline after one year of the pandemic in each participant with diabetes.
Number of patients with diabetes who have a higher BP (blood pressure) value (Change from baseline after 1 and 2 year of COVID 19 pandemic) | Baseline values - before the start of COVID 19 pandemic (1.9.2019 - 1.3.2020)- change from baseline after 1 year 1.4. - 31.7. 2020 and after 2 years (1.4.2021-31.7.2022)
  The investigators compare the value of blood pressure before the start of the COVID 19 pandemic and change from baseline after one year of the pandemic in each participant with diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vaclavik, Study Chair — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
Will be discussed.